CLINICAL TRIAL: NCT04866524
Title: Developmental Outcomes of Children Born Through Intracytoplasmic Sperm Injection (ICSI) Versus Conventional in Vitro Fertilization (IVF) in Couples With Non-male Factor Infertility
Brief Title: Child Follow-up in Women Treated With Conventional IVF or ICSI
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04/2021/MĐ-HĐĐĐ
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Conventional IVF, ICSI
MeSH Terms: interventions — Health Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICSI technique: In ICSI group, insemination will be performed by using ICSI, 3 - 4 hours after oocyte retrieval. OCCs will be stripped by using hyaluronidase. Only matured oocytes will be inseminated.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags
- Conventional IVF: In conventional IVF group, insemination will be performed by conventional IVF. Two hours after retrieval, collected OCCs will be inseminated for another 2 hours, at a concentration of 100,000 motile sperm/ml. Inseminated OCCs will be cultured overnight in culture medium.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags

INTERVENTIONS:
Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy to use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
Other: Physical development and General Health — Physical development and General health examination
Other: Developmental Red flags — Developmental Red flags Questionnaires

SUMMARY:
To compare the physical, mental and motor development of babies born from pregnancy using ICSI technique and and conventional IVF in non-male factor infertile couples. Based on our previous RCT (NCT03428919), the non-male factor couples were randomly assigned to IVF or ICSI, which leads to the similarity in characteristics of these two groups. Hence, the result of analyzing these offsprings would be preciously valuable.

DETAILED DESCRIPTION:
Over the past two decades, intracytoplasmic sperm injection (ICSI) indications have been extended and routinely applied to all cases of assisted reproductive techniques: unexplained infertility, poor-quality oocytes, low oocyte yeild, advanced marternal age, prior failed fertilization with conventional insemination, after in-vitro maturation of oocytes and for cases of cryopreserved oocytes (Practice Committees of the American Society for Reproductive Medicine, 2020). In 2004, fertilization using ICSI accounted for nearly 60% of all aspirations globally. In the Middle East, the number of ICSI cycles increased rapidly from 2000 (47.6%) to 2007 (65.2%), and reached 97.8% in the Middle East in 2007 (Ishihara et al, 2015). Another survey recorded in Europe in 2011, out of a total of 437,510 cycles of fresh embryo transfer, 68% of cycles were performed using ICSI techniques. In male infertility cases, the rate of implementation of ICSI increased from 76.3% to 93.3%. In particular, in cases of non-male-factor infertility, the incidence of ICSI also increased from 15.4% to 66.9%. From 2008-2012, of 494 907 treatment cycles, 74.6% used ICSI. In which, ICSI accounts for 92.9% of the cycle of male infertility and 64.5% of the cycle of non-male-factor infertility (Boulet, 2015).

However, ICSI is an invasive technique that bypasses the natural barriers of fertilization. This has led to concern about an increase in the incidence of anomalies in ICSI-born babies as this technique is increasingly being used in all cases of contraception. In contrast, there are studies that have also compared IVF with ICSI and show that in the ICSI cycle, the incidence of multiple pregnancies and low birth weight infants is lower than that of IVF, although there is no difference in infant survival between the two groups (Boulet et al, 2015).

In addition to the short-term outcomes, the investigators also have to consider the long-term maternal and neonatal outcomes. There is still not much evidence comparing the effects of the above methods, if any, on the psychomotor development in children.

Therefore, the investigators decide to conduct a study to compare the physical, mental and motor development of babies born from pregnancy using ICSI technique and and conventional IVF in non-male factor infertile couples.

ELIGIBILITY:
Inclusion Criteria:

* Live babies born from ICSI Versus Conventional IVF in Non-male Factor Couples (NCT03428919)
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died after the perinatal period.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Live babies born through intracytoplasmic sperm injection (ICSI) versus conventional in vitro fertilization (IVF) in couples with non-male factor infertility (NCT03428919)
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The number of patients having abnormal ASQ-3 scores in each aspect | Up to 66 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  Abnormal ASQ-3 score in an aspect = ASQ-3 score of 2 standard deviations below the mean of the aspect.

SECONDARY OUTCOMES:
Score of Communication | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Fine motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Problem solving | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Personal-Social | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
The rate of children who have at least one red flag sign | From 2 to 5.5 years after birth
  He or she has at least one red flag sign by age:
  From 12 to < 18 month-old:
  * Doesn't crawl
  * Can't stand when supported
  * Doesn't search for things that he/she sees the participants hide
  * Doesn't say single words ("baba", "mama"...)
  * Doesn't learn gestures like waving or shaking head
  * Doesn't point to things
  * Loses skills he/she once had
  From 18 to < 24 month-old:
  * Doesn't point to show things to others
  * Can't walk
  * Doesn't know what familiar things are for
  * Doesn't gain new words
  * Doesn't have at least 6 words
  * Doesn't notice or mind when a caregiver leaves or returns
  * Lose skills he once had
  From 24 to < 36 month-old:
  * Doesn't use 2-word phrases
  * Doesn't know what to do with common things, like a brush, spoon
  * Doesn't copy actions and words
  * Doesn't follow simple instructions
  * Doesn't walk steadily
  * Loses skills he/she once had
Duration of breast-feeding | Up to 24 months after birth
  Duration of breast-feeding
Infant age at which weaning starts | Up to 24 months after birth
  Infant age at which weaning starts
Name of diseases that lead to hospital admission | Up to 66 months after birth
  Name of diseases that lead to hospital admission
Weight | Through study completion, an average of 1.5 months
  Weight on the examination date
Height | Through study completion, an average of 1.5 months
  Height on the examination date

OTHER OUTCOMES:
The rate of long-term illness and chronic conditions | Up to 66 months after birth
  The rate of long-term illness and chronic conditions

CONTACTS AND LOCATIONS:
Overall Officials: Nghia A Nguyen, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen NA, Nguyen NT, Tran VTT, Vo TTM, Uong TS, Nguyen HT, Nguyen NT, Nguyen DL, Pham TD, Nguyen DTN, Ho TM, Vuong LN. Developmental outcomes of children born through ICSI versus conventional IVF (cIVF) in couples with non-male factor infertility. Hum Reprod. 2024 Jun 5:deae120. doi: 10.1093/humrep/deae120. Online ahead of print. PMID 38840410